CLINICAL TRIAL: NCT03637426
Title: Effect of Nano-hydroxyapatite and Low-level Laser Therapy on Dentin Hypersensitivity Control: Clinical, Randomized, Double-blind, Placebo-controlled Study
Brief Title: Effect of Nano-hydroxyapatite and LASER on Dentin Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Para (Other)
Responsible Party: Principal Investigator, Cecy Martins Silva, Clinical Professor, Universidade Federal do Para
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFPara-004
Record Dates: First submitted 2018-08-09; First posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Dentin Sensitivity
Keywords: nano-hydroxyapatite; Laser; desensitizing
MeSH Terms: conditions — Dentin Sensitivity | interventions — Lasers; Low-Level Light Therapy; nano-hydroxyapatite-collagen

STUDY DESIGN:
Intervention Model Description: Volunteers 18 to 50 years old with hypersensitive teeth were randomly assigned to 4 groups: GPLACEBO - positioning of the laser tip without light emission + placeo substance; GnHAP - positioning of the laser tip without light emission + nano-hydroxyapatite; GLASER - positioning of the laser tip with light emission + plcebo substance; GLASERnHAP - positioning by laser beam with light emission + nano-hydroxyapatite.
Who Masked: Participant, Investigator
Masking Description: For this double-blind study, the evaluator and the patient were blinded. Only one evaluator assessed pain sensitivity, who did not participate in the randomization process, and also did not know in which group the patient was. The volunteers evaluated in the experiment also were not aware of the treatment to which they were submitted. Both the Nano-P desensitizer and the placebo toothpaste have the same coloration and similar visual appearance. The desensitizers were placed in equal containers so that patients were not identified as to the application of the product.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GPLACEBO (Placebo Comparator): In this group, a toothpaste without addition of fluoride or any other desensitizing agent (Natural, Contente®, Uberlândia, MG, Brazil) was applied to hypersensitive dentine. The GPLACEBO volunteers were submitted to the application of placebo dentifrice on the vestibular surfaces of hypersensitive teeth with the aid of a Microbrush applicator (Microbrush, 3M ESPE, São Paulo, Brazil) for 10 minutes. Then, a rubber cup (Unid Microdont, São Paulo, SP, Brazil) mounted on a low speed handpiece (Dabi Atlante, Ribeirão Preto, SO, Brazil) was used to scrub the desensitizing gel on teeth for 20 seconds on each tooth.
  Interventions: Other: PLACEBO
- Gn-HAP (Experimental): In this group a desensitizing gel containing 20% of nano-hydroxyapatite, 9000 ppm of sodium fluoride and 5% of potassium nitrate (Desensibilize Nano P, FGM®, Joinville, SC, Brazil) was applied to the hypersensitive dentin. The GnHAP volunteers will be submitted to the application of Desensibilize Nano P on the vestibular surfaces of hypersensitive teeth with the aid of a Microbrush applicator (Microbrush, 3M ESPE, São Paulo, Brazil) for 10 minutes. Then, a rubber cup (Unid Microdont, São Paulo, SP, Brazil) mounted on a low speed handpiece (Dabi Atlante, Ribeirão Preto, SO, Brazil) was used to scrub the desensitizing gel on teeth for 20 seconds in each tooth, according to the manufacturer's specifications.
  Interventions: Other: nano-hydroxyapatite
- GLASER (Experimental): In this group, the diode laser with an active medium of Asauxa bauxite (Photon Lase III, DMC Equipamentos Ltda; São Carlos, SP, Brazil) was applied in hypersensitive dentine.
  GLASER received the laser application using the infrared light spectrum with wavelength of 808 nm with its active AsGaAl medium in two points of the vestibular face of the hypersensitive teeth. It was applied at each point 60 J / cm², for 16 seconds. The laser was applied in 2 sessions with a time interval of 24 hours.
  Interventions: Other: Laser
- GLASERnHAP (Experimental): In this group the laser + nano-hydroxyapatite was applied. The laser was used with light intensity medium Asauxa (Photon Lase III, DMC Equipamentos Ltda, São Carlos, SP, Brazil) and a gel containing 20% nanohydroxyapatite, 9000 ppm sodium fluoride 5% potassium nitrate (Desensibilize Nano P, FGM®, Joinville, SC, Brazil) in hypersensitive dentin. GLASERnHAP first named a laser application and then an application of nanohydroxyapatite according to the manufacturer's recommendations.
  Interventions: Other: Laser + nano-hydroxyapatite

INTERVENTIONS:
Other: Laser — GLASER received the laser application using the infrared light spectrum with wavelength of 808 nm with its active AsGaAl medium in two points of the vestibular face of the hypersensitive teeth. It was applied at each point 60 J / cm², for 16 seconds. The laser was applied in 2 sessions with a time interval of 24 hours.
  Other Names: Low level laser therapy
  Arms: GLASER
Other: nano-hydroxyapatite — The GnHAP volunteers were submitted to the application of Desensibilize Nano P on the vestibular surfaces of hypersensitive teeth with the aid of a Microbrush applicator (Microbrush, 3M ESPE, São Paulo, Brazil) for 10 minutes. Then, a rubber cup (Unid Microdont, São Paulo, SP, Brazil) mounted on a low speed handpiece (Dabi Atlante, Ribeirão Preto, SO, Brazil) was used to scrub the desensitizing gel on teeth for 20 seconds in each tooth, according to the manufacturer's specifications
  Other Names: dentin desensitization agent based on nano-hydroxyapatite
  Arms: Gn-HAP
Other: Laser + nano-hydroxyapatite — GLASERnHAP first received laser application and subsequently the application of nanohydroxyapatite according to the manufacturer's recommendations.
  Arms: GLASERnHAP
Other: PLACEBO — In this group, a toothpaste without addition of fluoride or any other desensitizing agent (Natural, Contente®, Uberlândia, MG, Brazil) was applied to hypersensitive dentine. The GPLACEBO volunteers were submitted to the application of placebo dentifrice on the vestibular surfaces of hypersensitive teeth with the aid of a Microbrush applicator (Microbrush, 3M ESPE, São Paulo, Brazil) for 10 minutes. Then, a rubber cup (Unid Microdont, São Paulo, SP, Brazil) mounted on a low speed handpiece (Dabi Atlante, Ribeirão Preto, SO, Brazil) was used to scrub the desensitizing gel on teeth for 20 seconds on each tooth.
  Arms: GPLACEBO

SUMMARY:
The aim of this study was to evaluate the effect of nanohydroxyapatite associated with low potency laser therapy in eliminating or reducing dentin hypersensitivity in a randomized placebo-controlled clinical trial. Volunteers 18 to 50 years old with hypersensitive teeth were randomized into 4 groups: GPLACEBO - positioning of the laser tip without light emission + placebo dentifrice; GnHAP - positioning of the laser tip without light emission + nano-hydroxyapatite; GLASER - laser tip positioning with light emission + placebo substance; GLASERnHAP - positioning by laser beam with light emission + nano-hydroxyapatite.

DETAILED DESCRIPTION:
GLASER received the laser application using the infrared light spectrum with wavelength of 808 nm with its active AsGaAl medium in two points of the vestibular face of the hypersensitive teeth. It was applied at each point 60 J / cm², for 16 seconds. The laser was applied in 2 sessions with a time interval of 24 hours. GLASERnHAP first received laser application and then the application of nanohydroxyapatite according to the manufacturer's recommendations. Before initiating laser therapy, the equipment was calibrated with a tester (MMOptics Ltda®, São Carlos, SP, Brazil).

The GnHAP volunteers were submitted to the application of Desensibilize Nano P on the vestibular surfaces of hypersensitive teeth with the aid of a Microbrush applicator (Microbrush, 3M ESPE, São Paulo, Brazil) for 10 minutes. Then, a rubber cup (Unid Microdont, São Paulo, SP, Brazil) mounted on a low speed handpiece (Dabi Atlante, Ribeirão Preto, SO, Brazil) was used to scrub the desensitizing gel on teeth for 20 seconds in each tooth, according to the manufacturer's specifications. GPLACEBO followed the same protocol used in Gn-HAP. In addition to the desensitization treatment, all GnHAP and GPLACEBO volunteers received the positioning of the laser tip to mimic the light emission produced in GLASER and GLASERnHAP. The noise emitted by the laser device during mimicry was simulated through the sound reproduction of a smartphone application (HD Voice Recorder - iPhone 6s, Apple®, Cupertino, California, USA).

ELIGIBILITY:
Inclusion criteria:

- The presence of at least one hypersensitive tooth;

Exclusion criteria:

* patients with systemic diseases;
* patients with pulpitis;
* patients with carious lesions;
* patients with defective restorations;
* patients with cleft enamel;
* patients with active periodontal disease;
* patients with analgesic medication;
* patients with pregnant or lactating women
* patients who have received professional desensitizing treatment in the last three months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-08-03 (Actual)

PRIMARY OUTCOMES:
Pain intensity change | up to 2 months
  Self reported intensity dentin sensitivity before and after desensitizing treatment. Each item is scored 1-10 (0-no pain and 10- pain as bad as can be)

CONTACTS AND LOCATIONS:
Overall Officials: Cecy M Silva, pHD, Principal Investigator — Federal University of Para
Locations (1):
- Federal University of Pará, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: Undecided